CLINICAL TRIAL: NCT04819932
Title: An Open-label, Randomized, 2x2 Crossover Study to Compare the Pharmacokinetics and Safety Following Administration of DWJ1451 and Co-administration of DWC202008 and DWC202009 in Healthy Volunteers
Brief Title: Pharmacokinetics and Safety of DWJ1451 in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWJ1451102
Record Dates: First submitted 2021-01-27; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group1 (Experimental): subject take DWC202008 and DWC2020091 on a fasted condition, and after wash out period, take DWJ1451 with on a fasted condition
  Interventions: Drug: DWJ1451
- group2 (Experimental): subject take DWJ1451 on a fasted condition, and after wash out period, take DWC202008 and DWC202009 with on a fasted condition
  Interventions: Drug: DWJ1451

INTERVENTIONS:
Drug: DWJ1451 — DWC202008 DWC202009

SUMMARY:
Amlodipine, olmesartan, total ezetimibe, rosuvastatin AUCt, Cmax

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 55 years
* Healthy Adult

Exclusion Criteria:

* Non-Healthy

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-03-13 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-04-02 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of DWJ1451:AUC0-t | 0 - 72 hours after dosing
  Area under the plasma xonxentration-time curve from time 0 to t
Pharmacokinetic parameter of DWJ1451:Cmax | 0 - 72 hours after dosing
  Maximum plasma drug concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea